CLINICAL TRIAL: NCT03536611
Title: A Randomized Study Comparing Dabigatran Etexilate Versus Warfarin in Chinese Patients With Nonvalvular Atrial Fibrillation Who Undergo Percutaneous Coronary Intervention With Stenting (DES)
Brief Title: Dabigatran Versus Warfarin With NVAF Who Undergo PCI
Acronym: COACH-AF-PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Northern Hospital (Other)
Collaborators: Beijing Anzhen Hospital (Other); Second Affiliated Hospital of Third Military Medical University (Other)
Responsible Party: Principal Investigator, Han Yaling, Director, clinical professor, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYNH-K201813
Record Dates: First submitted 2018-04-25; First posted 2018-05-24 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
Keywords: dabigatran; warfarin; non-valve atrial fibrillation; percutaneous coronary intervention
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dabigatran (Experimental): dabigatran etexilate 110 mg bid + aspirin 100 mg qd + clopidogrel 75 mg qd for 1 month followed by dabigatran 110mg bid + clopidogrel 75mg/d for at least 5 months
  Interventions: Drug: dabigatran
- warfarin (Active Comparator): warfarin (according to clinical routine monitoring of INR, maintain the therapeutic range at 2.0-3.0) + aspirin 100 mg qd + clopidogrel 75 mg qd for 1 month followed by warfarin + clopidogrel 75mg/d for at least 5 months
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: dabigatran — dabigatran etexilate 110 mg bid + aspirin 100 mg qd + clopidogrel 75 mg qd for 1 month followed by dabigatran 110mg bid + clopidogrel 75mg/d for at least 5 months
  Arms: dabigatran
Drug: warfarin — warfarin (according to clinical routine monitoring of INR, maintain the therapeutic range at 2.0-3.0) + aspirin 100 mg qd + clopidogrel 75 mg qd for 1 month followed by warfarin + clopidogrel 75mg/d for at least 5 months
  Arms: warfarin

SUMMARY:
This study is to compare the efficacy and safety of dabigatran ethidium b.i.d.+ clopidogrel + ASA [100 mg q.d. *1 month] and warfarin + clopidogrel + ASA [100 mg, q.d.*1 month] in Chinese NVAF patients undergoing PCI with stenting (elective or due to ACS).

DETAILED DESCRIPTION:
This is an open-label, multi-center, randomized, controlled, prospective study.The object of this study is to compare the safety and efficacy of dabigatran etexilate combined with dual anti-platelet therapy versus warfarin combined with dual anti-platelet therapy in Chinese patients with nonvalvular atrial fibrillation who undergo percutaneous coronary intervention.

The subjects are randomized into study group and control group using central randomization for open-label dosing:(1) Study group: dabigatran etexilate 110 mg bid + aspirin 100 mg qd + clopidogrel 75 mg qd. Aspirin is withdrawn 1 month later;(2) Control group: warfarin (according to clinical routine monitoring of INR, maintain the therapeutic rang at 2.0-3.0) + aspirin 100 mg qd + clopidogrel 75 mg qd. Aspirin is withdrawn 1 month later;All patients should receive the study medication for 6 month.

Primary endpoint:Time to the first occurrence of BARC-defined (grade 2-5) clinically relevant bleeding.

Key secondary endpoint:Time to the first occurrence of net clinical adverse events. Net clinical adverse event is composed of major cardiovascular and cerebrovascular adverse events (all death, recurrent myocardial infarction, ischemia-induced revascularization of the target vessel, or stroke/systemic embolism) or BARC-defined (grade 2-5) clinically relevant bleeding.

Secondary endpoints:1) Major cardiovascular and cerebrovascular adverse events 2) Major bleeding or clinically relevant non-major bleeding (ISTH definition) 3) Major bleeding (ISTH definition) 4) Any bleeding event (BARC-defined grade 1-5) 5) Clinically relevant bleeding (BARC-defined grade 2-5) 6) Bleeding (BARC-defined grade 3-5)

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Patients with non-secondary (e.g., pericarditis, hyperthyroidism, recent surgery, etc.) nonvalvular atrial fibrillation requiring long-term anticoagulant treatment;
3. Patients who have PCI indications and coronary heart disease that was successfully treated with drug-eluting stenting (DES);
4. Patients who sign the informed consent form. -

Exclusion Criteria:

1. Patients with mechanical or biological heart valve prosthesis;
2. Patients proposed to undergo left atrial appendage occlusion or atrial fibrillation radiofrequency ablation
3. Cardiogenic shock during current hospitalization;
4. Patients who have used fibrinolytic agents within 24 hours of randomization that, in the opinion of the Investigator, will put the patient at high risk of bleeding;
5. Stroke within 1 month prior to screening visit;
6. Patients, who in the opinion of the Investigator, have had major surgery within the month prior to screening;
7. Patient has received an organ transplant or is on a waiting list for an organ transplant;
8. History of intraocular, spinal, retroperitoneal or a traumatic intra-articular bleeding unless the causative factor has been permanently eliminated or repaired (e.g. by surgery);
9. Gastrointestinal (GI) haemorrhage within one month prior to screening, unless, in the opinion of the Investigator, the cause has been permanently eliminated (e.g. by surgery);
10. Major bleeding episode (reduction in the haemoglobin level of at least 2 g/dL, transfusion of at least two units of blood, or symptomatic bleeding in a critical area or organ) including life-threatening bleeding episode (symptomatic intracranial bleeding, bleeding with a decrease in the haemoglobin level of at least 5 g/dL or bleeding requiring transfusion of at least 4 units of blood or inotropic agents or necessitating surgery) in one month prior to screening visit;
11. Haemorrhagic disorder or bleeding diathesis (e.g. von Willebrand disease, haemophilia A or B or other hereditary bleeding disorder, history of spontaneous intra-articular bleeding, history of prolonged bleeding after surgery/intervention);
12. Anaemia (haemoglobin <10 g/dL) or thrombocytopenia including heparin-induced thrombocytopenia (platelet count <100×109/L) at screening (Visit 1);
13. Severe renal impairment (estimated CrCl calculated by Cockcroft-Gault equation) <30 mL/min at screening;
14. Active liver disease as indicated by at least one of the following:

    * Prior and persistent alanine aminotransferase (ALT) or Aspartate transaminase (AST) or alkaline phosphatase (AP) >3 upper limit of normal (ULN);

      * Known active hepatitis C; ③Known active hepatitis B; ④Known active hepatitis A;
15. Recent malignancy or radiation therapy (≤6 months) unless, in the opinion of the Investigator, the estimated life expectancy is greater than 36 months;
16. Need for continued treatment with systemic ketoconazole, itraconazole, posaconazole, cyclosporine, tacrolimus, dronedarone, rifampicin, phenytoin, carbamazepine, or any cytotoxic/myelosuppressive therapy;
17. Patients who, in the Investigator's opinion, need continuous treatment with Non-Steroidal Anti-Inflammatory Drugs (NSAIDs);
18. Patients with a known allergy to dabigatran etexilate or to the excipients used for the capsule of the drug
19. Patients with a known allergy to warfarin tablets or to the excipients
20. Patients who, in the Investigator's opinion, should not be treated with OAC;
21. Patients with a contraindication to clopidogrel, or ASA
22. Pre-menopausal women (last menstruation ≤1 year prior to screening) who experienced any of the following conditions:

    * Are pregnant or breast feeding; ②Are pregnant surgically sterile; ③Are of child bearing potential and not practising two acceptable methods of birth control, or do not plan to continue practising an acceptable method of birth control throughout the trial. (Acceptable methods of birth control are oral or parenteral (patch, injection, implant) hormonal contraception which has been used continuously for at least one month prior to the first dose of study medication, intrauterine device or intrauterine system, double-barrier method of contraception (condom and occlusive cap or condom and spermicidal agent), male sterilization and complete sexual abstinence (if acceptable by local authorities)). Periodic abstinence is not an acceptable method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
clinically relevant bleeding | 24 months
  Time to the first occurrence of BARC-defined (grade 2-5) clinically relevant bleeding.

SECONDARY OUTCOMES:
Time to the first occurrence of major cardiovascular and cerebrovascular adverse events | 24 months
  Time to the first occurrence of net clinical adverse events. Net clinical adverse event is composed of major cardiovascular and cerebrovascular adverse events (all death, recurrent myocardial infarction, ischemia-induced revascularization of the target vessel, or stroke/systemic embolism) or BARC-defined (grade 2-5) clinically relevant bleeding.

OTHER OUTCOMES:
other events | 24 months
  1. Major cardiovascular and cerebrovascular adverse events
  2. Major bleeding or clinically relevant non-major bleeding (ISTH definition)
  3. Major bleeding (ISTH definition)
  4. Any bleeding event (BARC-defined grade 1-5)
  5. Clinically relevant bleeding (BARC-defined grade 2-5)
  6. Bleeding (BARC-defined grade 3-5)

CONTACTS AND LOCATIONS:
Overall Officials: zulu Wang, PhD, Principal Investigator — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liang M, Jin J, Zhao R, Li H, Chen S, Liu L, Xu P, Wang W, Cheng X, Chen X, Tao L, Zhang Q, Yang M, Zeng C, Li L, Zheng Y, Chen H, Guo J, Zhong Z, Bi Y, Cheng B, Zhou Y, Wang H, Zhang Y, Qiu M, Zhang Q, Zhang P, Zhang J, Wang Z, Li Y, Han Y. Dabigatran-based versus warfarin-based triple antithrombotic regimen with a 1-month intensification after coronary stenting in patients with nonvalvular atrial fibrillation (COACH-AF PCI). BMC Med. 2025 Nov 18;23(1):643. doi: 10.1186/s12916-025-04477-1. PMID 41254594